CLINICAL TRIAL: NCT01108757
Title: Prevention of Catheter-Associated Urinary Tract Infections in Patients Undergoing Incontinence and Reconstructive Pelvic Surgery: A Randomized Controlled Trial
Brief Title: Prevention of Catheter-Associated Urinary Tract Infection in Incontinence and Reconstructive Pelvic Surgery Patients
Acronym: PRECAUTION
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unfeasible because of low accrual
Sponsor: The Cleveland Clinic (Other)
Collaborators: American Urogynecologic Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 10-125
Record Dates: First submitted 2010-04-21; First posted 2010-04-22 (Estimated); Results first posted 2017-10-18 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Catheter-Associated Urinary Tract Infection
Keywords: catheter; urinary tract infection
MeSH Terms: conditions — Urinary Tract Infections | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug (Experimental)
  Interventions: Drug: Bactrim
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Bactrim — Bactrim DS BID for 3 days
  Arms: Drug
Other: Placebo — Corn starch capsules
  Arms: Placebo

SUMMARY:
The study will assess the risk of catheter associated urinary tract infection in women undergoing incontinence or reconstructive pelvic surgery. Women will be given an antibiotic or placebo at the time of catheter removal. The investigators hypothesize that prophylactic antibiotics will reduce the rate of infection.

ELIGIBILITY:
Inclusion Criteria:

* Requires catheterization >24h hours following incontinence or pelvic reconstructive surgery

Exclusion Criteria:

* Receipt of antibiotics for either prophylaxis or treatment of a known infection during the postoperative hospitalization
* Allergy to sulfonamides or trimethoprim
* Non-English speaking
* Pregnancy
* Breast feeding
* Severe renal impairment (creatinine clearance <30)
* Patients taking dofetilide, methenamine, procaine, warfarin, procainamide, methotrexate.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2010-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D Barber, MD MHS, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 52 subjects were recruited.
Period: Overall Study
Arm/Group | Drug | Placebo
Started | 26 | 26
Completed | 26 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Drug: Bactrim: Bactrim DS BID for 3 days
  Demographics data by group not available as this study was discontinued in 2013. Currently randomization data not available for reassessment.
- Total: Total of all reporting groups
Arm/Group | Drug | Placebo | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Customized [Mean (Standard Deviation); unit: years]
  Mean Age | 60 (12.9) | 58 (13.0) | 59 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 52
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 26 | 52
Body mass index [Mean (Standard Deviation); unit: kg/m^2] — Body mass index (BMI) measured as kg/m^2
  kg/m^2 | 25.8 (2.7) | 27.2 (4.3) | 26.5 (3.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Urinary Tract Infection
Description: Urinary tract infection diagnosis was obtained after confirmation with urine culture microbiology report. Infection was defined as >100,000 colony forming units/mL
Time Frame: 7 days following catheter removal
Population: Study terminated early.
Measure: Count of Participants; unit: Participants
Arm/Group | Drug | Placebo
Number analyzed (Participants) | 26 | 26
Participants | 6 | 6

ADVERSE EVENTS:
Time Frame: 3-years while patients were in treatment and follow-up
Arm/Group | Drug | Placebo
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No